CLINICAL TRIAL: NCT00520611
Title: Evaluating the Effectiveness of Financial Incentives in Promoting Weight Loss Among Obese Individuals.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: William and Flora Hewlett Foundation (Other); USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00985
Record Dates: First submitted 2007-08-22; First posted 2007-08-24 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2010-01

CONDITIONS: Obesity
Keywords: Obesity; Weight Loss; Financial Incentives; Lottery; Deposit
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lottery (Active Comparator): Participants are entered into daily lotteries to win $10 or $100 every day their weight is at or below daily targets.
  Interventions: Behavioral: Financial Incentives
- Deposit (Active Comparator): Participants receive $3/day if they are at or below their daily weight goals, plus have opportunity to deposit up to $3/day of their own money, which is then matched 1:1 every day they are at or below their daily weight goals.
  Interventions: Behavioral: Financial Incentives
- Control (No Intervention): Participants would receive usual care from their providers and have monthly weigh ins.

INTERVENTIONS:
Behavioral: Financial Incentives — Participants call in their weight on daily basis. Participants must report under their daily targets to qualify for entry into lottery. Call-in weights are verified at monthly weigh-ins.
  Arms: Lottery
Behavioral: Financial Incentives — Participants call in their weight on daily basis. Participants must report under their daily targets to qualify to receive daily incentive. Call-in weights are verified at monthly weigh-ins.
  Arms: Deposit

SUMMARY:
Obesity is a major cause of premature aging and the second leading cause of preventable mortality in the United States, accounting for approximately 110,000 deaths per year. Financial incentives have been effective in modifying a number of health behaviors but they have rarely been applied to weight loss, and to the best of our knowledge never to weight loss by low-SES obese veterans.

We propose testing two different approaches to using financial incentives to encourage weight loss. In the first, we build on previous work showing the effectiveness of 'deposit contracts', in which subjects are given the opportunity to put their own money at risk if they do not lose weight. In this incentive condition, subjects receive a direct payment conditional on daily weight loss, and an optional additional payment based on their own contributions to the deposit contract. We will match their contribution 1:1 to make the option of depositing their own money attractive to this predominantly low SES population. In the second approach we build on our own prior work using lotteries to promote drug adherence. In this incentive condition, participants are entered into a daily lottery, and receive any payoffs they earn from the lottery only if they stay on track with their weight-loss goal. Given their popularity in the general population, lotteries hold the promise of providing a cost-effective means of motivating weight loss and making efforts to lose weight more salient to obese patients.

DETAILED DESCRIPTION:
Fifty-seven obese patients at the Philadelphia VAMC (BMI between 30-40) will be randomly assigned to one of three conditions: weight monitoring only (WM), deposit contract incentive (DC$+WM), or lottery-based incentive (L$+WM). Exclusion criteria for the study will be minimal to maximize generalizability, focusing only on exclusions that may make participation unfeasible or unsafe (myocardial infarction within 6 months; uncontrolled hypertension, defined as BP>170 mm Hg systolic or BP>110 mm Hg diastolic; metastatic cancer, self-report of 6 or more alcoholic beverages per day; schizophrenia; severe depression; active substance abuse; inability to read or severe cognitive deficits that would preclude ability to read consent form or fill out surveys). Patients with severe depression will be referred for treatment and considered ineligible until effectively treated. This exclusion is appropriate because those who are severely depressed are too ill to undertake weight reduction and because weight loss is often a symptom of severe depression. Subjects will also be asked how interested they are in losing weight (5 point scale, ranging from extremely uninterested to extremely interested, minimum score of 3 for inclusion). Subjects will be required to be between ages 30-70, as weight loss may be more difficult and less beneficial in the elderly. No other exclusions will be applied, as we aim to make the study as generalizable as possible. Initial screening of BMI's and comorbidities will be done using the VALOR data system at CHERP. Subjects who on paper meet criteria will then be sent letters and asked to call us if interested. The remaining eligibility criteria will be assessed over the phone, and subjects who meet the criteria will be invited for an in-person intake visit.

At the initial intake visit, study procedures will be explained, and staff will create a linear graph depicting the course of weight loss required to lose 16 pounds over the course of 16 weeks (see figure). Subjects who provide written consent to participate will be randomized to one of the 3 arms at this visit. Participants randomized to one of the two incentive arms will be informed of the incentive plan (described in detail below). Physiologic measurements will be limited to weight and height which will be measured by our staff. To minimize fluctuations in weight due to diurnal variation, subjects will be asked to commit to having all morning appointments (e.g. between 8 and 1 pm) for both intake and f/u visits if possible. For those who cannot come in mornings, they will be asked to commit to coming in at approximately the same time in the afternoon for intake and f/u visits (e.g. between 2 and 4 pm). As soon as possible, following the intake visit, all participants will have a one-on-one consultation with a dietician (Kelly McBride) in which diet and exercise will be discussed. During this session, participants will receive guidance on strategies for weight loss.

Following this consultation, participants will be asked to return to PVAMC to see the coordinator at CHERP once a month for each of four consecutive months to: be weighed (all participants), receive any payment they have earned (DC$+WM) or (L$+WM), and complete a follow-up questionnaire. Subjects will be instructed to drink only one 8 ounce glass of liquid and have a small breakfast and/or lunch (Examples of a small breakfast would be 2 slices of whole grain toast with jelly or one serving of a whole grain cereal with skim milk or a piece of fruit and glass of skim milk. Light lunch could include any of the ones listed above, or a broth based soup or half of a turkey sandwich or half of a peanut butter) prior to coming in for follow-up visits. To compensate subjects for their time and trouble, all participants will receive a financial incentive each time they attend a monthly weigh-in, regardless of whether or not they have attained their monthly weight loss goal. Subjects will also receive a financial incentive for attending the initial intake visit and a financial incentive for attending their appointment with the dietician (Kelly McBride) and for coming to a f/u weigh in at 3 months after the incentives for weight loss cease. Those in the two incentives conditions will be provided with daily feedback, as described below. All such messages will be transmitted by text -enabled pagers that we will provide for the duration of the study for this purpose.

Subjects will be asked to measure their weight each morning upon awakening, after urinating, but before eating or drinking and to transmit it to the study administrator by telephone (by leaving a message). We will provide scales that are accurate to 0.1 pounds to each subject for use for the duration of the study. We will tell participants at entry into the study that the scale is theirs to keep if they remain enrolled in the study for the duration but that they will be asked to return them if they drop out of the study before then. These scales will be calibrated initially to match the weights recorded by the scale used at CHERP.

As mentioned above, there will be two different financial incentive conditions that we will be testing, both of which have a strong conceptual basis and for which there is suggestive evidence in the literature that these could be effective approaches to help obese patients lose weight.

Patients randomized to the lottery financial incentives arm will be eligible for a daily lottery prize with an expected value of $3/day (a rough estimate of the savings per day to a health plan from reducing the incidence of type 2 diabetes and other consequences of obesity by achieving weight loss of 10-20 lbs) only if, prior to the lottery being resolved, they have reported a weight at or below their desired weight loss trajectory (see figure). The lottery is tailored both to provide infrequent large payoffs (a 1 in 100 chance at a $100 reward) and frequent small payoffs (a 1 in 5 chance at a $10 reward). This is because lottery players are motivated by both a forward looking element (fixation on large $ amounts) and a backward looking element - how often did I win.

The lottery is designed such that, each day, subjects who send their early morning weights will receive rapid feedback about whether they won, and non-adherent subjects will receive feedback about whether they would have won had they been adherent. Subjects will be asked to choose a 2-digit number upon entry into the study, e.g. "27". Each morning subjects will be asked to call in to report their weight from that morning. A two digit random number will be generated for each day. If the last digit includes either a "2" or "7" (which has approximately a 1 in 5 chance), and the subject reported a weight that was at or below their target weight for that day, they would be eligible to win $10. If the number is "27" (a 1 in 100 chance) they would win $100. Information on whether they won would be transmitted to them each day, via text message, so that they receive this feedback immediately. If a subject does not report their weight that morning (by 12pm) or reports a weight that is above the target weight (with an allowance for the inaccuracy of the scale), they will be informed that they would have won the lottery that day had they been below target. We believe that a desire to avoid the regret associated with not winning, but learning that one would have won had one been adherent, will powerfully motivate subjects to adhere - beyond what one might anticipate based only on the expected value of the rewards. Moreover, this effect will probably strengthen with experience - i.e., after a given subject has experienced the remorse of failing to obtain rewards that they would have received if they had been adherent. Subjects who achieve a 20 pounds or more weight loss over the 16 weeks will be eligible for a one-time bonus of at least $50.

Because the above daily weights are all self-reported, we will inform patients that they will only receive the calculated amount they are due if their weight at their monthly weigh-in is at or below their target weight (typically a 4 pound weight loss over 1 month). A 0.2 pound differential will be allowed between the office scale reading and the participant's reported weight at the time of their monthly visit to account for 0.1 pound scale variances on either the office or take home scales (e.g. if a subject loses 3.8 instead of 4.0 pounds per the office scale, they will receive their full incentive). These payments would be provided using the "Authorization and Invoice for Medical and Hospital Services Form" that allows participants to be paid directly through VA Agent Cashier.

Deposit contract financial incentive ($+WM) participants will be paid a base amount corresponding to $3 for each day they are on track toward losing 16 pounds of weight by the end of the 16-week study. Specifically, they receive this payment for every day that their weight is at or below the ideal threshold line (see figure). In addition, these participants will be given the opportunity to contribute between $0-$3 per day of their own funds, refundable at the end of the month only if they have met or exceeded their monthly weight loss goal. As an incentive for participants to contribute to deposit contracts, we will match their money 1:1. Thus, participants in this condition have the opportunity to earn as much as $9 per day ($3 base payment plus their $3 plus our $3 match). Participants will decide at the beginning of each month how much, if any, they wish to deposit for the upcoming month. They can therefore change the amount of their deposit contracts from month to month. Any deposit contract money that is forfeited by participants because they do not lose a sufficient amount of weight will be contributed to a pool of money that will be divided equally among all subjects who lose 20 pounds or more over the 16 weeks. The size of this bonus will be not less than $50, with any shortfall to be made up by study funds. Because not all subjects will complete the study at the same time we will give each subject who is eligible for this bonus $50 at the final follow-up visit. If the eventual amount ends up being more, we will mail them a money order or the "Authorization and Invoice for Medical and Hospital Services Form" to make up the difference.

Participants will be asked to self-monitor their weight on a daily basis and to transmit it to the central office by phone. Each morning before eating or drinking and after urinating, participants will be asked to a) weigh themselves in their pajamas, b) record their weights, and c) transmit their weight to the central office before 12 noon. To maintain comparability between the lottery and deposit contract groups, every afternoon, participants will receive a text message telling them whether they are below their threshold weight for payment and, if they are, how much they have received; if they are not at or below their threshold weight, how much they would have received if they had been. At their monthly weigh-in, participants will be given a report that captures how their report weights compare to the ideal weight loss trajectory sketched in the initial consultation session and giving them information on how much they will be paid if these weights are accurate, as well as how much they would have received if they had stayed on target.

The daily monitoring provides participants with a constant reminder of their weight loss goals. This frequency was chosen based on the finding that people tend to adopt a narrow (daily) frame of reference to diets, "rededicating" themselves to it at the start of each day. The daily weigh-ins are designed to reduce binge eating by making participants constantly "accountable" for their weight. The monthly feedback provides encouragement and a symbolic reward for slow and steady weight loss.

Falsification of weights will be minimized because patients will only get paid the amounts identified in the weekly reports if the degree of weight loss recorded at the monthly weigh-ins done by our coordinator are consistent with their self reports.

A key aspect of the weight loss trajectory is that it can be reset at monthly intervals. This feature is critical in the likely event that a person falls short of attaining a monthly weight loss goal. Disheartened at the prospect of having to lose double the weight in order to get "back on track" by the end of the next month, such a person might drop out of the study. To avoid this problem, each person who has not reached the weight loss for the previous month will be given the opportunity for a "fresh start." The overall weight loss goal will stay the same, however, the slope of the trajectory will adjust (i.e. steepen) such that the participant need not "binge diet" following a month of poor weight loss performance (see "Fresh start trajectory" in figure, which assumes the subject lost 2 lbs. instead of 4 lbs. in first month). Keeping the overall weight loss goal constant makes the procedure fair for those participants who maintain the ideal trajectory, while adjusting the slope of the weight loss line allows for subjects who have occasional slip-ups to stay engaged and get back on track.

Our standard approach to receiving information from subjects will involve subjects calling us by telephone. We will not require subjects to have access to a home computer and electronic mail.

Weight Monitoring only participants (control group) will be given the goal of losing 16 pounds in 16 weeks but will receive usual care only, e.g. care provided by their regular clinical providers. They will not be given any financial incentive to lose the weight. They will be asked to come for a monthly f/u visit and weigh in, but will not receive any communications between these visits from the study coordinator.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 30-40;
* Age between 30-70;
* At least moderately interested in losing weight (Self-reported 3,4, or 5 on 5 point scale)

Exclusion Criteria:

* Unstable medical conditions that would likely prevent the subject from completing the study;
* Myocardial infarction within 6 months;
* Uncontrolled hypertension, defined as BP>170 mm Hg systolic or BP>110 mm Hg diastolic;
* Metastatic cancer;
* Self-report of 6 or more alcoholic beverages per day;
* Severe depression;
* Active substance abuse;
* Schizophrenia
* Inability to read or severe cognitive deficits that would preclude ability to read consent form or fill out surveys.
* Baseline participation in other weight loss programs.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2007-06; Primary Completion 2008-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Mean weight loss will be greater in both experimental groups compared to the control group by the end of 16 weeks | 4 months

SECONDARY OUTCOMES:
Use the difference in weight loss measured at 16 weeks to project the long-term cost-effectiveness if weight loss is sustained | 4 Months

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Volpp, MD, PhD, Principal Investigator — Univesity of Pennsylvania; George Loewenstein, PhD, Study Director — Carnegie Mellon University; Leslie John, PhD cand., Study Director — Carnegie Mellon University
Locations (1):
- Center for Health Equity Research and Promotion, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Volpp KG, John LK, Troxel AB, Norton L, Fassbender J, Loewenstein G. Financial incentive-based approaches for weight loss: a randomized trial. JAMA. 2008 Dec 10;300(22):2631-7. doi: 10.1001/jama.2008.804. PMID 19066383